CLINICAL TRIAL: NCT01899040
Title: A Non-Invasive Neuromodulation Device for Treatment of Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNS-MIG-01
Record Dates: First submitted 2013-06-29; First posted 2013-07-15 (Estimated); Results first posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Migraine Headache, Episodic
Keywords: neuromodulation; migraine headache; CVS
MeSH Terms: conditions — Migraine Disorders; Recurrence

STUDY DESIGN:
Intervention Model Description: The study was designed with two arms - active and placebo. The devices for the first 20 placebo-randomized participants were found to be partially active. Therefore, the fully placebo arm was separated into placebo and partially active placebo. Only the active and placebo arms were followed (and outcomes posted) for effectiveness. All (active, placebo, and partially active) were followed and outcomes posted for safety.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active device (Active Comparator): A standardized active neuromodulation waveform will be used for all active Device patients at all Study sites. The Device will be used twice daily.
  Interventions: Device: neuromodulation for episodic migraine headache
- placebo device (Placebo Comparator): A standardized placebo neuromodulation waveform will be used for all placebo Device patients at all Study sites. The Device will be used twice daily.
  Interventions: Device: neuromodulation for episodic migraine headache

INTERVENTIONS:
Device: neuromodulation for episodic migraine headache

SUMMARY:
This is a randomized, blinded study designed to assess the efficacy of a portable, non-invasive neuromodulation system for the treatment of episodic migraine headaches.

DETAILED DESCRIPTION:
This is a multi-center, triple-blinded, placebo-controlled, randomized pivotal trial evaluating the adjunctive prophylactic treatment of episodic migraine headache using a caloric vestibular stimulation (CVS) device developed by Scion NeuroStim, LLC (SNS). This study has been reviewed by the FDA and is categorized as posing NSR (nonsignificant risk).

ELIGIBILITY:
INCLUSION CRITERIA:

* The patient must have been diagnosed with episodic Migraine Headache at least 6 months prior to entering into the Study, consistent with the International Headache Classification of Headache Disorders-II (ICHD-II) guidelines.
* The patient must have a history of at least three consecutive months of stable Migraine Headaches prior to entering the Study. The patients will not have had changes in medication usage for the three Months leading up to the Study, nor will they introduce new medications during the Study period. Patients will satisfy these criteria: On a Monthly basis, at least four, and not more than a total of fourteen (4-14), Headache Days (Pain Score between one and ten) of which between four and nine (4-14) are Migraine Headache Days
* The patient must not have failed on more than two classes of properly administered prophylactic pharmaceutical therapies for migraine headache. The patient may be on a single migraine prophylactic as long as the dosage has not been altered within 3 months of starting the study and the dosage must not be altered for the duration of the study.
* The Investigator must have confidence in the patient's ability to reliably use the Experimental Device and promptly complete the Daily Headache Diary forms. The Daily Headache Diary will be completed from the beginning of the Pre-Treatment Baseline Period through the end of the Pivotal Study.

EXCLUSION CRITERIA:

Individuals who:

* are pregnant
* have a history of cardiovascular disease
* work night shifts
* have been diagnosed with vestibular migraine
* have been diagnosed with migraine with aura
* have menstrual migraine exclusively
* have been diagnosed with post-traumatic migraine
* have a history of unstable mood disorder or unstable anxiety disorder
* use a hearing aid
* have a cochlear implant
* have chronic tinnitus
* have temporomandibular joint (TMJ) disease
* have been diagnosed with traumatic brain injury (TBI)
* have been diagnosed with neurological disease other than Headaches
* have a diagnosed vestibular dysfunction
* abuse alcohol or other drugs
* are experiencing medication overuse Headaches (individuals with respect to whom the Investigator is concerned that analgesic abuse is involved based on the ICHD-II guidelines).
* are younger than 18 years or older than 65 years
* have had eye surgery within the previous three months or ear surgery within the previous six months
* have active ear infections or a perforated tympanic membrane
* have participated in another clinical trial within the last 30 days or are currently enrolled in another clinical trial
* are using Botox treatments for migraines
* Though not excluded, patients taking anti-histamines or anti-nausea drugs will be encouraged not to take such medications within four hours prior to using the Device. The Investigator should review other medications taken by the patient with properties that mimic anti-nausea or anti-dizziness drugs as these may reduce responsiveness to stimulation. Such medications should also be avoided within four hours prior to a treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesco Rogers, MD, Study Director — Scion NeuroStim
Locations (6):
- United States (5):
  - Naval Medical Center, San Diego, California
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Carolina Headache Institute, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
- Kent University, Canterbury, Kent, United Kingdom

REFERENCES:
- [Derived] Wilkinson D, Ade KK, Rogers LL, Attix DK, Kuchibhatla M, Slade MD, Smith LL, Poynter KP, Laskowitz DT, Freeman MC, Hoffer ME, Saper JR, Scott DL, Sakel M, Calhoun AH, Black RD. Preventing Episodic Migraine With Caloric Vestibular Stimulation: A Randomized Controlled Trial. Headache. 2017 Jul;57(7):1065-1087. doi: 10.1111/head.13120. Epub 2017 Jun 27. PMID 28656612

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Device: A standardized, active tvCVS neuromodulation waveform treatment delivered by a device used twice daily for all active Device patients at all Study sites.
- Placebo Device (Inactive Device): A standardized, fully-inactive placebo tvCVS neuromodulation waveform treatment delivered twice daily by the study device was used for this group at all Study sites.
- Placebo Device (Partially Active): The description of this treatment is a standardized partially-active neuromodulation waveform delivered twice daily was used for the first 20 participants randomized to the placebo group at all Study sites.
  While the participants in this group were supposed to have received a fully-inactive waveform, their devices were found to be delivering an unintended partially-active treatment. This was discovered well after the study had begun. As their results did not represent use of a true (i.e., fully inactive) device, these participants were separated from the main placebo group and followed for safety only for the duration of the study.
Period: Overall Study
Arm/Group | Active Device | Placebo Device (Inactive Device) | Placebo Device (Partially Active)
Started | 50 | 30 | 20
Completed | 42 | 22 | 17
Not Completed | 8 | 8 | 3
Not completed — Randomized in error | 0 | 1 | 1
Not completed — Adverse Event | 3 | 1 | 2
Not completed — Unspecified reasons | 4 | 4 | 0
Not completed — Compliance issues | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis populations include the fifty (50) participants who were randomized BID Active, the thirty (30) participants who were randomized to BID Placebo and received BID Placebo (fully inactive), and the twenty (20) who were randomized to BID Placebo BUT received Partially-Active devices.
Groups:
- BID Active: Participants (episodic migraineurs) self-administered twice-daily active treatments for 12 weeks
  The Device delivered a standardized, active tvCVS neuromodulation waveform twice-daily to all active Device patients at all Study sites.
- BID Inactive Placebo: Participants (episodic migraineurs) self-administered twice-daily inactive/sham treatments for 12 weeks
  The Device delivered a standardized, placebo (no power to the earpieces) tvCVS neuromodulation waveform twice-daily to all inactive placebo Device patients at all Study sites.
- BID Partially-Active Placebo: Participants (episodic migraineurs) self-administered twice-daily partially active treatments for 12 weeks
  The description of this treatment is a standardized partially-active neuromodulation waveform delivered twice daily was used for the first 20 participants randomized to the placebo group at all Study sites.
  While the participants in this group were supposed to have received a fully-inactive waveform, their devices were found to be delivering an unintended partially-active treatment. This was discovered well after the study had begun. As their results did not represent use of a true (i.e., fully inactive) device, these participants were separated from the main placebo group and followed for safety only for the duration of the study.
- Total: Total of all reporting groups
Arm/Group | BID Active | BID Inactive Placebo | BID Partially-Active Placebo | Total
Number analyzed (Participants) | 50 | 30 | 20 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Only participants that had data for this baseline measure were included in the analysis. Two (2) inactive placebo participants did not have baseline population for this baseline measure.
  Years
    number analyzed (Participants) | 50 | 28 | 20 | 98
    (all) | 44.0 (11.1) | 40.7 (12.4) | 42.3 (8.6) | 42.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 28 | 17 | 89
  Male | 6 | 2 | 3 | 11
Disease Duration [Mean (Standard Deviation); unit: Years] — Population: Only participants with data for this baseline analysis measure were included in this analysis. Disease duration was not collected for two(2) BID Active, one (1) BID Placebo, and three (3) BID Partially-Active Placebo participants.
  Years
    number analyzed (Participants) | 48 | 29 | 17 | 94
    (all) | 24.5 (12.4) | 20.8 (10.5) | 17.6 (8.4) | 22.1 (11.4)
Years of Education [Mean (Standard Deviation); unit: Years] — Population: Only participants with data reported for this baseline measure are included in the analysis. Education data was not collected for four (4) BID Active and three (3) BID Placebo participants.
  Years
    number analyzed (Participants) | 46 | 27 | 20 | 93
    (all) | 16.2 (2.6) | 16.2 (2.6) | 15.3 (2.5) | 16.0 (2.6)
Baseline migraine days [Mean (Standard Deviation); unit: days] — The number of days with a migraine headache reported during the 28-day baseline period, based on a headache diary Population: Only participants with data reported for this baseline measure are included in the analysis. Data is missing for this baseline measure due to the original headache diaries being either inaccessible or not completed by the participants at the time of the study.
  days
    number analyzed (Participants) | 39 | 19 | 16 | 74
    (all) | 7.7 (2.5) | 6.9 (2.9) | 8.3 (2.5) | 7.6 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Monthly Migraine Headache Days
Description: Change in the average total number of Monthly Migraine Headache Days (number of days in the month that a participant experienced a migraine) after 3 months of treatment comparable to the pre-device use Baseline Period of 1 month, as reported in a headache diary. Negative number indicated improvement (a reduction in the average number of migraine headache days experienced per month).
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria, received either placebo (completely inactive) or fully active devices, and completed this outcome effectiveness measures were included in the overall number of participants analyzed for this outcome. Additional missing data comes from participants not being fully compliant with headache diary.
Measure: Mean (Standard Deviation); unit: migraine days
Groups:
- BID Active Device: A standardized, active tvCVS neuromodulation waveform treatment delivered by a device used twice daily for all active Device patients at all Study sites.
- BID Placebo (Fully Inactive Device): A standardized, fully-inactive placebo tvCVS neuromodulation waveform treatment delivered twice daily by the study device was used for this group at all Study sites.
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device)
Number analyzed (Participants) | 38 | 19
migraine days | -3.5 (0.6) | -1.1 (0.6)

2. Secondary Outcome: Number of Monthly Migraine Headache Days (Reduction by by 50% or More)
Description: Number of participants that experienced a reduction of 50% or more in Monthly Migraine Headache Days (total days during a month on which a migraine occurred) during the third month of device use as compared with their pre-device use Baseline Period.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria & received either placebo (completely inactive) or fully active devices and completed primary and secondary outcome effectiveness measures were included in the overall number of participants analyzed for this outcome.
  For both Active and Placebo, all participants with baseline and third month of data were included in analysis. Additional missing data comes from participants not being fully compliant with headache diary.
Measure: Count of Participants; unit: Participants
Groups:
- Fully Inactive Placebo Device: A standardized placebo neuromodulation waveform will be used for all placebo Device patients at all Study sites. The Device will be used twice daily.
Arm/Group | Active Device | Fully Inactive Placebo Device
Number analyzed (Participants) | 38 | 19
Participants | 20 | 6

3. Secondary Outcome: Total Monthly Headache Pain Score
Description: After three months of Device use, the average Total Monthly Headache Pain Score compared to the average derived from the Pre-use Baseline Period (1 month). This is calculated by adding the cumulative maximum pain scores for all days the subject had a headache, as noted as the maximum daily headache pain score on a scale of 1 (lowest pain)-10 (highest pain) for each headache day as reported by the subject in their daily headache diary. Each month was counted as 28 days. Therefore, the total possible score for each month was 28-280. A negative number indicates a reduction in pain score.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria, received either active or placebo (completely inactive) treatments, and completed this effectiveness measure were included in the overall number of participants analyzed for this outcome.
  Additional missing data comes from participants not being fully compliant with headache diary.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Device | Fully Inactive Placebo Device
Number analyzed (Participants) | 38 | 19
score on a scale | -19.3 (3.6) | -10.3 (3.4)

4. Secondary Outcome: (Safety Measure) Mood and Cognition - Change in Beck Depression Index Score
Description: A patient's Pre-device use Baseline Period mood score from the Beck Depression Index is compared with those at the end of the 3 month Device use period. The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression, with each of the 21 items, rated on a 4-point scale (0-3). The total scores rage from 0-63. The higher the score the more depressed. Mood scores are assessed for: decline, no change, or an improvement. A negative score indicates improvement in mood.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria and completed baseline and month 3 for this measure were included in the overall number of participants analyzed for this outcome. As this is a safety measure, all (active, placebo, and partially active) participants were followed and outcomes presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BID Placebo (Partially Active): A standardized, partially-active placebo tvCVS neuromodulation waveform treatment delivered twice daily by the study device was used for this group at all Study sites.
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device) | BID Placebo (Partially Active)
Number analyzed (Participants) | 40 | 22 | 17
score on a scale | -0.7 (0.4) | -0.9 (0.7) | -0.9 (1.4)

5. Secondary Outcome: (Safety Measure) Dizziness: Verify the Absence of Change in Material Dizziness (Berg Balance)
Description: The purpose of this study endpoint is to verify, using the Berg Balance test, the absence of change in material dizziness (with the associated risk of falls) as a consequence of using the Device. The test consists of 14 balance- related tasks ranging from standing up from a sitting position to standing on one foot. Each task is graded from 0 - 4, and the final measure is the sum from all elements of the Test: • 41-56 = low risk of fall • 21-40 = medium risk of fall • 0-20 = high risk of fall. Possible scores range from 0-56. Scores of zero indicate no change in balance.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria and completed this measure were included in the overall number of participants analyzed for this outcome. As this is a safety measure, active, placebo, and partially active groups were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BID Placebo (Partially-active): A standardized, partially-active placebo tvCVS neuromodulation waveform treatment delivered twice daily by the study device was used for this group at all Study sites.
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device) | BID Placebo (Partially-active)
Number analyzed (Participants) | 42 | 22 | 17
score on a scale | 0.0 (0.0) | 0.0 (0.0) | 0.3 (0.4)

6. Secondary Outcome: (Safety Measure) Mood and Cognition - Change in Digit Symbol Coding Cognitive Speed
Description: A patient's Pre-use Baseline Period cognitive speed scores, using the Digit Symbol Coding assessment, will be compared with those at the end of the Device use period. The Digit-Symbol Subtest of the WAIS-III, is a timed pencil-and-paper task that measures processing speed and visual-motor coordination. It involves matching symbols to numbers using a key, with the goal of completing as many correct matches as possible within a 120-second time limit. The number of correct matches completed is counted. The lowest possible count is 0 (zero correct matches). The higher the number of correct matches completed, the better the cognitive speed of the participant. Cognitive speed will be assessed for: a decline, no change, or an improvement. A positive number indicates improvement.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria and completed this safety measure were included in the overall number of participants analyzed for this outcome. As this was a safety measure, active, placebo and partially active groups were followed and results presented.
Measure: Mean (Standard Deviation); unit: tasks completed
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device) | BID Placebo (Partially-active)
Number analyzed (Participants) | 40 | 22 | 17
tasks completed | 7.1 (1.9) | 5.0 (1.9) | 7.4 (2.9)

7. Secondary Outcome: (Safety Measure) Mood and Cognition Measure - Change in Short Term Memory Test Scores
Description: A patient's Pre-use Baseline Period memory scores, using Short Term memory test (an old/new paradigm for face recognition) are compared with those at the end of the 3-month Device use period. This assessment was created by the study Neuropsychologist where participants were shown faces at baseline then shown another set which included a subset then had seen before and had to say if they had seen them before later during the visit (to test short term memory). Scores range from 0-10. Higher scores indicate better short term memory. Memory scores were assessed for: a decline, no change, or an improvement from baseline to the end of treatment month 3. A negative score indicates improvement.
Time Frame: after 84 days of Device use
Population: Only participants who were confirmed to meet eligibility criteria and completed this outcome measure were included in the overall number of participants analyzed for this outcome. As this was a safety measure, all (active, placebo, and partially active) participants with baseline and third month of data were included in analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BID Active Device: A standardized active neuromodulation waveform will be used for all active Device patients at all Study sites. The Device will be used twice daily.
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device) | BID Placebo (Partially-active)
Number analyzed (Participants) | 40 | 22 | 17
score on a scale | -1.0 (1.0) | -1.9 (1.5) | 1.0 (1.5)

8. Secondary Outcome: Average of Monthly Treated Headaches (Acute Anti-migraine Prescription Drug Intake)
Description: This measures counts the number of times abortive medications are taken. The baseline count is subtracted from the third month count. A negative number indicates a reduction in abortive medications used. The greater the negative number, the more reduced the use of abortive medications.
Time Frame: after 84 days of device use
Population: Only participants who were confirmed to meet eligibility criteria and had baseline and month 3 data for this outcome were included in the overall number of participants analyzed for this outcome. As this is an effectiveness measure, only Active and Placebo (fully inactive) participants were followed and included in analysis. Additional missing data comes from participants not being fully compliant with headache diary.
Measure: Mean (Standard Deviation); unit: # acute antimigraine medication intakes
Arm/Group | BID Active Device | BID Placebo (Fully Inactive Device)
Number analyzed (Participants) | 38 | 19
# acute antimigraine medication intakes | -3.5 (0.6) | -1.8 (0.8)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: clinicaltrials.gov terms were used.
Groups:
- Placebo Device (Fully-inactive Device): A standardized, fully-inactive placebo tvCVS neuromodulation waveform treatment delivered twice daily by the study device was used for this group at all Study sites.
- Placebo Device (Partially Active Device): The description of this treatment is a standardized partially-active neuromodulation waveform delivered twice daily was used for the first 20 participants randomized to the placebo group at all Study sites.
  While the participants in this group were supposed to have received a fully-inactive waveform, their devices were found to be delivering an unintended partially-active treatment. This was discovered well after the study had begun. As their results did not represent use of a true (i.e., fully inactive) device, these participants were separated from the main placebo group and followed for only safety (adverse events and safety outcome measures) for the duration of the study.
Arm/Group | Active Device | Placebo Device (Fully-inactive Device) | Placebo Device (Partially Active Device)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 14/50 | 7/30 | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Device (N=50) | Placebo Device (Fully-inactive Device) (N=30) | Placebo Device (Partially Active Device) (N=20)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Sinus Infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 3 (5) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Cold (Infections and infestations) | 5 (5) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
The devices of the first 20 placebo-randomized participants were found to be delivering a partially active treatment. Not yet distributed devices were corrected to ensure they were fully inactive and were supplied to all other placebo-randomized participants thereafter. 2 participants were found to have not met the criteria after inclusion into the study. These results weren't included in the primary/some secondary outcome analyses, as they artificially inflated the effectiveness of the device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT01899040/Prot_SAP_000.pdf